CLINICAL TRIAL: NCT00958347
Title: Omnifit Hydroxylapatite (HA) Hip Outcomes Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to lagging follow-up
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01/04
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-07

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omnifit HA Hip Stem (Other): Participants underwent total hip replacement surgery using the Omnifit HA Hip Stem.
  Interventions: Device: Omnifit HA Hip Stem

INTERVENTIONS:
Device: Omnifit HA Hip Stem — Total Hip Replacement with Omnifit HA Hip Stem

SUMMARY:
The purpose of this study was to obtain up to 25 year post-operative data on the Omnifit Hydroxylapatite (HA) Hip System in support of the hypothesis that it is a satisfactory system for reducing implant loosening, permitting tissue bonding onto the hydroxylapatite surfaces of the implant and providing a safe, efficient, and well-functioning hip in a wide spectrum of clinical circumstances.

ELIGIBILITY:
Inclusion Criteria:

For use as a universal hip replacement:

* Acute femoral neck fracture.
* Non-union of femoral head and neck fractures.
* Aseptic necrosis of the femoral head.
* Osteoarthritis, rheumatoid arthritis, or post-traumatic arthritis of the hip with minimal acetabular involvement or distortion.
* Salvage of failed total hip arthroplasty.

For use as a total hip replacement:

* Severely disabled joints resulting from painful osteoarthritis, rheumatoid arthritis, or post-traumatic arthritis.
* Revision of previous unsuccessful femoral head replacement, cup arthroplasty, or other procedure.

Exclusion Criteria:

* Active infection in or near the hip joint.
* Pathological bone conditions which would significantly compromise the ability to carry physiologic stress levels and for which bone grafting would be inappropriate (i.e. severe osteoporosis, Paget's Disease, renal osteodystrophy, etc.).
* Neuro-muscular disorders in which the potentially adverse effects on prosthesis function are not outweighed by the benefits to be gained by the patient from usage of the implant.
* Mental disorders which would compromise essential patient post-operative care.
* Skeletal immaturity.
* Extreme obesity.
* Significant probability that patient could not return for required follow-up evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 1987-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Capello, MD, Study Chair — Indiana University School of Medicine; William Jaffe, MD, Principal Investigator — Hospital for Joint Disease/ Orthopaedic Institute; Rudolph Geesink, MD, Principal Investigator — Trialbureau Orthopedics; James D'Antonio, MD, Study Chair — Sewickley Valley Hospital
Locations (4):
- United States (3):
  - Indiana University Medical Center, Indianapolis, Indiana
  - Hospital for Joint Disease/ Orthopaedic Institute, New York, New York
  - Sewickley Valley Hospital, Moon Township, Pennsylvania
- Trialbureau Orthopedics, Maastricht, Netherlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 226 participants = 262 hips
Period: Overall Study
Arm/Group | Omnifit HA Hip Stem
Started | 226
Completed | 0 (11 revisions total, one was a bilateral participant with the other hip counted as not completed.)
Not Completed | 226
Not completed — Death | 43
Not completed — Withdrawal by Subject | 23
Not completed — Lost to Follow-up | 15
Not completed — revision/removal | 10
Not completed — study termination | 135

BASELINE CHARACTERISTICS:
Arm/Group | Omnifit HA Hip Stem
Number analyzed (Participants) | 226
Age, Continuous [Mean (Standard Deviation); unit: years] — For bilateral total hip replacement participants, the age at the time of the initial hip replacement surgery is used.
  years | 51.55 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 113

OUTCOME MEASURES:

1. Primary Outcome: Patients Will be Evaluated for Pain, Functional Level, and Clinical Complications Utilizing the Harris Hip Score.
Time Frame: 25 Years Post-Operatively
Population: The study was closed and no subjects reached the 25 year postoperative endpoint.
Arm/Group | Omnifit HA Hip Stem
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 22 years
Description: Elective procedures are not included. These may include: non-study total knee/hip replacements/revisions, rotator cuff repairs, carpal tunnel releases, cataract & intra-ocular procedures, bunion procedures, total shoulder repairs, laminectomies, microdiscectomies, breast reductions, cervical spine fusions, & mid-foot/flat-foot surgeries.
Arm/Group | Omnifit HA Hip Stem
Serious Adverse Events (participants affected / at risk) | 104/226
Other Adverse Events (participants affected / at risk) | 70/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omnifit HA Hip Stem (N=226)
Non-operative Site Cardiac Disorders (Cardiac disorders) | 13 (13)
Non-operative Site Gastrointestinal Disorders (Gastrointestinal disorders) | 1 (1)
Non-operative Site Infections and Infestations (Infections and infestations) | 2 (2)
Operative Site Infection and Infestation (Infections and infestations) | 2 (3)
Non-operative Site Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 9 (9)
Operative Site Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 81 (122)
Non-Operative Site Neoplasms Benign,Malignant,and Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Non-operative Site Renal and Urinary Disorders (Renal and urinary disorders) | 1 (1)
Operative Site Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 1 (1)
Non-operative Site Vascular Disorders (Vascular disorders) | 9 (9)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omnifit HA Hip Stem (N=226)
Non-operative Site Musculoskeletal and Connective Tissue Disorder (Musculoskeletal and connective tissue disorders) | 19 (26)
Operative Site Musculoskeletal and Connective Tissue Disorder (Musculoskeletal and connective tissue disorders) | 59 (75)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For 7 years from and after termination date of the agreement, prior to submission for publication of abstracts, manuscripts, presentations or other communications describing the results of any aspect of the Study ("Manuscript"), You and the Institution shall send Stryker Orthopaedics a copy of the Manuscript to be submitted, and allow Stryker Orthopaedics sixty (60) days from the date of receipt to review the Manuscript.